CLINICAL TRIAL: NCT03716349
Title: Esthetic Outcomes of a Newly Developed Dental Composite and Adhesive System: a Randomized Clinical Trial
Brief Title: Esthetics of Dental Composite and Adhesive System
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Erica Teixeira (Other)
Collaborators: Tokuyama Dental Corporation (Unknown)
Responsible Party: Sponsor-Investigator, Erica Teixeira, Principal Investigator, University of Iowa
Organization: University of Iowa (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 201809844
Record Dates: First submitted 2018-10-01; First posted 2018-10-23 (Actual); Last update posted 2025-06-05 (Actual); Status verified 2025-05

CONDITIONS: Cavities of Teeth
MeSH Terms: conditions — Dental Caries | interventions — Anesthetics, Local; Rubber Dams; Consent Forms; Patient Health Questionnaire; X-Rays; Diagnosis, Oral

STUDY DESIGN:
Intervention Model Description: Simple randomization will be used for assignment of the treatment groups. Randomization: Two restorations will be placed in each subject, one using system A and one using system B.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: The statistician will prepare a randomization list of A-B and B-A pairs to be applied sequentially as subjects receive restorations. The first system listed in the randomization pair will be placed on first tooth (#4-#13), and the second system on 2nd tooth (#4-#13). The random sequence will be individually placed in opaque, consecutively numbered and sealed envelopes, which should be opened by the operator immediately before the intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- System A (Experimental): Tokuyama Universal Bond (TUB) single component self-etching 1-step adhesive system w/Tokyuama supra-nanofilled dental composite (ECM) (Tokuyama Dental Corp., Japan), informed consent signed, release of medical information signed, oral exam, health Questionnaire completed and/or updated, xray obtained if needed, pulp vitality testing, Tooth shade determination, photos of teeth, local and/or topical anesthetic applied as necessary, rubber dam isolation, tooth surface cleaned, cavity preparation performed as usual for caries removal, Enamel margins beveled, infinite invisible margins created, adhesive systems applied, dental composite placed, shade selection using Easy Shade 5. Light curing, restoration will be contoured and polished. teeth assessment, clinical assessment
  Interventions: Diagnostic Test: Pulp vitality testing; Other: Photos; Drug: local and/or topical anesthetic; Device: rubber dam; Other: tooth surface cleaned; Procedure: enamel margins; Procedure: Adhesive Systems; Procedure: cavity preparation; Other: Shade selection using Easy Shade 5; Procedure: Light Curing; Procedure: Contoured and polished; Other: Consent; Other: Health Questionnaire; Radiation: xray; Other: Release of medical information signed; Other: Oral Exam; Other: Teeth Assessment; Other: Clinical Assessment; Device: Tokuyama Universal Bond
- System B (Active Comparator): ScotchBond Universal one-step adhesive system with Filtek Supreme Ultra™, nanofilled dental composite (3M) will randomly be applied to the other tooth informed consent signed, release of medical information signed, oral exam, health Questionnaire completed and/or updated, xray obtained if needed, pulp vitality testing, Tooth shade determination, photos of teeth, local and/or topical anesthetic applied as necessary, rubber dam isolation, tooth surface cleaned, cavity preparation performed as usual for caries removal, Enamel margins beveled, infinite invisible margins created, adhesive systems applied, dental composite placed, shade selection using Easy Shade 5. Light curing, restoration will be contoured and polished. teeth assessment and clinical assessment at periodic timepoints.
  Interventions: Diagnostic Test: Pulp vitality testing; Other: Photos; Drug: local and/or topical anesthetic; Device: rubber dam; Other: tooth surface cleaned; Procedure: enamel margins; Procedure: Adhesive Systems; Procedure: cavity preparation; Other: Shade selection using Easy Shade 5; Procedure: Light Curing; Procedure: Contoured and polished; Other: Consent; Other: Health Questionnaire; Radiation: xray; Other: Release of medical information signed; Other: Oral Exam; Other: Teeth Assessment; Other: Clinical Assessment; Device: ScotchBond

INTERVENTIONS:
Diagnostic Test: Pulp vitality testing — each tooth will be tested to determine if the pulp of the tooth responds to cold
Other: Photos — Photos of teeth (Photos will be taken with a DSLR camera settings will be determined with optimal settings) and captured periodically throughout the study. Photographs will be made of the cavity preparation. Photographs will be made post-operatively
Drug: local and/or topical anesthetic — Local and/or topical anesthetic will be applied as necessary to the teeth or gingiva
Device: rubber dam — The area will be isolated with rubber dam isolation
Other: tooth surface cleaned — The tooth surface will be cleaned with flour of pumice on a prophy cup only, cavity preparation will be performed as usual for caries removal.
Procedure: enamel margins — Enamel margins will be beveled with a long flame diamond bur (8863.314.012 Komet) at 45 degrees to the external tooth surface to achieve the desired bevel length. Along with the use of the diamond bur, infinite invisible margins will be created by contouring and smoothing with a dark orange Sof-LexTM extra-thin contouring and polishing disc (3M).
Procedure: Adhesive Systems — Adhesive systems will be applied according to manufacturer's instructions and selective etching of the enamel will be performed. The dental composite will be incrementally placed using a two- layer or one-layer technique based on the cavity size and light-cured (detailed adhesive instruction sheet will be chairside for reference)
Procedure: cavity preparation — The technique to be used will be determined by the size of the final cavity preparation. For small preparations a one-layer technique will be used. No backing material is necessary for the Tokuyama system, Filtek Supreme Ultra will be determined by manufacturer's wheel. A two-layer technique will be used for a large cavity preparation. Large cavity preparation is defined as being 4mm in length or more and/or at least 2mm in depth.
Other: Shade selection using Easy Shade 5 — A1 (shade determined by Easy Shade 5), ECM-001/Backing material, A1E/A2D (shade will be selected by shade wheel) A4 (shade determined by Easy shade5), ECM-001/Backing material, A3E/A6D (shade will be selected by shade wheel
Procedure: Light Curing — A Valo Grand curing unit (Ultradent) with an exitant irradiance with no less than 500 and no greater than 1500 mW/cm2 as measured with MARC Light Collector will be used in standard mode to deliver the required radiant exposure J/cm2 for adhesive and dental composite increments.
Procedure: Contoured and polished — The restoration will be contoured and polished with - Long flame diamond bur (8863.314.012 Komet), Sof-Lex Medium (orange) Contouring and Polishing Discs (3M), Green Jiffy cup pre-polisher (Ultradent Products, Inc.), Blue and grey silicone points composite polisher gloss plus finisher (Kerr Hawe)
Other: Consent — The consent form will be signed, copy will be provided to the patient
Other: Health Questionnaire — The health questionnaire will be completed at initial visit and updated at each follow-up visit
Radiation: xray — When necessary a radiograph (xray) will be obtained
Other: Release of medical information signed — The release of medical information form will be signed
Other: Oral Exam — An Oral Exam will be completed
Other: Teeth Assessment — The teeth assessment by subject will be completed using the Visual Analog Scale (VAS) and Verbal Rating Scale (VRS) at the follow-up visits 1 month after restoration, 1 year, 2 years and 3 years post restoration.
Other: Clinical Assessment — A clinical assessment will be completed by the evaluators
Device: Tokuyama Universal Bond — Tokuyama Universal Bond (TUB) single component self-etching 1-step adhesive system with Tokyuama supra-nanofilled dental composite (ECM) (Tokuyama Dental Corp., Japan)
  Arms: System A
Device: ScotchBond — Scotch Bond Universal one-step adhesive system with Filtek Supreme Ultra™, nanofilled dental composite (3M)
  Arms: System B

SUMMARY:
To compare a newly developed filling composite to a current filling composite system. Two restorations will be placed in each subject, one using system A and one using system B. The first system listed in the randomization pair will be placed on first tooth (#4-#13), and the second system on 2nd tooth (#4-#13). The same three researchers will be responsible for placement of all the restorations.

DETAILED DESCRIPTION:
The aim of this (12-month; 36-month; 60-month) randomized controlled clinical trial is to evaluate and compare the esthetic outcomes and patient satisfaction of a simplified newly developed dental composite system (system A)for the esthetic region to a nanohybrid composite system (Filtek Supreme Ultra-system B) placed in class III, IV and V lesions. Even though dental composite systems have been used extensively for the anterior region, clinicians face challenges with shade selection and longevity of the material over the years. This new system has been developed to improve the esthetic outcomes and patient satisfaction by enhancing the blending capability of the material.

Dental composite systems have been used for 50 years as state of art materials to restore the anterior region. Significant development has occurred regarding the composition and structure of dental composites, improving the longevity of these restorations; however, clinicians are faced with the challenge of selecting the most adequate shade and restorative technique to reproduce missing tooth structure.

Depending on the size of the cavity preparation, a single layer of material or multiple layers might be needed to reproduce dentin and enamel. Different dental composite systems offer multiple body, dentin, and enamel shades. Therefore, clinicians are faced with the challenge of recreating nature using this material. Different devices, such as spectrophotometers have been introduced on the market for shade selection. However, one of the most important aspects when placing anterior composites is the esthetic outcome based on the patient's assessment. Therefore, this study will evaluate the esthetic outcomes of a simplified and a conventional dental composite system based on the provider's and patient's assessment.

ELIGIBILITY:
Inclusion Criteria:

* Sensible tooth -responds to cold or electric pulp testing (done at screening)
* Patient 18years of age or old
* Current radiograph available (done at screening as needed)
* A pair of the same type of restorations needed in the anterior esthetic/facial region (tooth #4-#13).

Exclusion Criteria:

* Fewer than 20 teeth
* Advanced untreated periodontal disease or recent periodontal surgery
* Rampant uncontrolled caries activity
* Bruxism or clenching and visible wear facets on the occlusal surface
* Undergoing or in need of TMJ therapy
* Known allergy to methacrylate-based materials or product ingredients
* History of poor dental visit attendance
* Not available for recall for at least 3 years
* Fractured or visibly cracked tooth
* Poor oral hygiene
* Sensitive tooth or currently using desensitizing treatments, pastes or medicaments
* Pregnant
* Abutment teeth for prostheses
* Teeth considered for restoration are non-vital, have had root canal therapy or been pulp capped
* Teeth or supporting structures with any symptomatic pathology or extensive caries lesion
* Individual supervised by PI or supervised by member of research team
* Individual subordinate to the PI or subordinate to any member of the research team
* Student or trainee under the direction of the PI or under the direction of a member of the research team

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Patient satisfaction of the restoration appearance (esthetics) VAS | 3 years and 5 years
  Patient satisfaction-VAS (Visual Analog Scale of 0-10 with 0 poor and 10 excellent result)

SECONDARY OUTCOMES:
Patient satisfaction of the restoration appearance (esthetics) VRS | 3 years and 5 years
  Patient satisfaction- VRS (Verbal Rating Scale - very satisfied to not at all satisfied)
Percent success of the restoration according to the esthetic appearance | baseline, 1 year, 3 years, 5 years
  Esthetic outcomes using the World Dental Federation instrument (FDI criteria- 5-likert scale criteria 1-best to 5 worst score) measured by the clinician's evaluators
Percent success of the restoration according to biological aspects | baseline, 1 year, 3 years, 5 years
  using the World Dental Federation instrument (FDI criteria- 5-likert scale criteria 1-best to 5 worst score) by the clinician's evaluator
Percent success of the restoration according to functional aspects | baseline, 1 year, 3 years, 5 years
  using the World Dental Federation instrument (FDI criteria- 5-likert scale criteria 1-best to 5 worst score) by the clinician's evaluator

CONTACTS AND LOCATIONS:
Overall Officials: Erica Teixeira, DDS, MS, PhD, Principal Investigator — University of Iowa College of Dentistry
Locations (1):
- University of Iowa, Iowa City, Iowa, United States

IPD SHARING:
Plan to Share IPD: No